CLINICAL TRIAL: NCT02110706
Title: B Cell Targeted Treatment In Myasthenia Gravis (BeatMG): A Phase II Trial of Rituximab In Myasthenia Gravis
Brief Title: BeatMG: Phase II Trial of Rituximab In Myasthenia Gravis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 1401013253-0; 1U01NS084495-01A1 (NIH); U01NS077179-01 (NIH); U01NS077352 (NIH)
Record Dates: First submitted 2014-04-07; First posted 2014-04-10 (Estimated); Results first posted 2018-10-02 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; Rituximab; SNOMED code 31839002
MeSH Terms: conditions — Myasthenia Gravis | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The placebo group will receive a vehicle control infusion
  Interventions: Drug: Placebo
- Rituximab (Experimental): Intervention (rituximab): The treatment group will receive a total of two cycles of rituximab separated by 6 months. Each cycle is defined as one infusion (375mg/m2 IV) per week for four consecutive weeks
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Intervention (rituximab): The treatment group will receive a total of two cycles of rituximab separated by 6 months. Each cycle is defined as one infusion (375mg/m2 IV) per week for four consecutive weeks
  Arms: Rituximab
Drug: Placebo — The placebo group will receive a vehicle control infusion
  Arms: Placebo

SUMMARY:
The specific primary objective of this study is to determine whether rituximab is a safe and beneficial therapeutic for Myasthenia Gravis (MG) that warrants further study in a phase III efficacy trial.

DETAILED DESCRIPTION:
Investigators plan on conducting a multicenter randomized, double-blind, placebo controlled Phase II clinical trial utilizing a futility design. The study would include acetylcholine receptor (AChR) antibody positive generalized MG subjects. This study also presents a unique opportunity to study both drug and disease mechanisms because unlike many other autoimmune diseases in which rituximab has been used, MG affords the investigation of antigen-specific components that participate in the immunopathology of the disease, namely autoantibodies, autoantibody-producing B cells, and antigen-specific T cells. This work will further our understanding of MG immunopathology and it represents the first step toward gaining a more complete understanding of the immune mechanisms underlying treatment of MG with rituximab leading to new ways to treat the disease.

The specific aim of this study is to determine whether rituximab is a safe and effective treatment for subjects with MG.

The SNOMED code for MG is 31839002.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 21 to 90 years old
2. Subjects must have generalized MG, defined as MGFA clinical classification grades 2 (mild), 3 (moderate), or 4 (severe, but not intubated) at the time of screening/randomization.
3. Elevated AChR antibody titer
4. Subject's signs and symptoms should not be better explained by another disease process.
5. Subjects must be on a stable standard immunosuppressive regimen:

   1. Prednisone only: Prednisone dose must be at least 15mg/day (or the equivalent on alternate days), and the dose of prednisone must have been stable for at least 4 weeks (28 days) prior to the baseline visit.
   2. Prednisone plus another immunosuppressive therapy (IST). Immunosuppressive therapies other than prednisone, specifically azathioprine, mycophenolate mofetil, cyclosporine, tacrolimus or methotrexate, are permitted, but the dose must have been stable for at least 6 months prior to the baseline visit.

   (Note: The prednisone dose must be stable as defined in the prednisone only group. The IST dose must remain stable throughout the course of the study).
6. Subjects must be willing to complete the study and return for follow-up visits.
7. No history of thymoma, tumor, infection, or interstitial lung disease on chest CT, MRI, or chest x-ray. Note: Chest x-ray will be completed at screening to look of interstitial lung disease. A chest CT or MRI to evaluate for thymoma must be completed as part of prescreening.
8. Able and willing to give written informed consent and comply with the requirements of the study protocol.
9. Subjects must be able to give written informed consent before participating in this study. A copy of the signed consent must be kept in the subject's medical record.
10. Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.

Exclusion Criteria:

1. A history of chronic degenerative, psychiatric, or neurologic disorder other than MG that can produce weakness or fatigue.
2. Other major chronic or debilitating illnesses within six months prior to study entry.
3. Female subjects who are premenopausal and are:

   1. pregnant on the basis of a serum pregnancy test,
   2. breast-feeding, or
   3. not using an effective method of double barrier (1 hormonal plus 1 barrier method or 2 simultaneous barrier methods) or birth control (birth control pills, male condom, female condom, intrauterine device, Norplant, tubal ligation, or other sterilization procedures).
4. Altered levels of consciousness, dementia, or abnormal mental status.
5. Thymectomy in the previous six months.
6. Subjects who have been medicated with immunosuppressive drugs not listed in inclusion #5 within the last 8 weeks (56 days) prior to the baseline visit
7. Subjects who have been medicated with an immunosuppressive agent such as azathioprine, mycophenolate mofetil, cyclosporine, tacrolimus or methotrexate, that is withdrawn within 8 weeks (56 days) of the Baseline Visit.
8. Subjects who have received IVIg or PLEX treatment within the last 4 weeks (28 days) prior to the baseline visit.
9. Unstable dose or a stable dose of > 480 mg/day of pyridostigmine in 2 weeks prior to screening visit.
10. Daily use of non-steroidal anti-inflammatory drugs (NSAIDs).
11. History of renal or hepatic insufficiency or elevated liver enzymes (AST or ALT >2.5 x Upper Limit of Normal).
12. History of bone marrow hypoplasia, leucopenia, thrombocytopenia, significant anemia, clinical or laboratory evidence of immunodeficiency syndromes.
13. Forced Vital Capacity (FVC) <50% of percent predicted.

    General Safety & Laboratory Exclusion Criteria
14. ANC < 1.5 x 103 cells/microliter
15. Hemoglobin: < 8.0 gm/dL
16. Platelets: < 100,000/mm
17. Positive Hepatitis B or C serology (Hep B surface antigen and Hep C antibody)
18. History of positive HIV (HIV conducted during screening if applicable)
19. Treatment with any investigational agent within 4 weeks of screening or 5 half-lives of the investigational drug (whichever is longer)
20. Receipt of a live vaccine within 4 weeks prior to randomization
21. Previous treatment with rituximab (MabThera® / Rituxan®)
22. Previous treatment with natalizumab (Tysabri®)
23. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
24. History of recurrent significant infection or history of recurrent bacterial infections
25. Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
26. Unstable steroid dose in the past 4 weeks (28 days)
27. Lack of peripheral venous access
28. History of drug, alcohol, or chemical abuse within 6 months prior to screening
29. Concomitant malignancies or previous malignancies, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or prostate.
30. History of psychiatric disorder that would interfere with normal participation in this protocol
31. Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
32. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications
33. Subjects that do not record daily prednisone doses for at least 28 days before the Baseline Visit, or subjects whose prednisone dose varies by ≥6mg/day on average.
34. Prednisone dose of more than 100 mg/day (or 200 mg over a two day period).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-05; Primary Completion 2017-07 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Nowak, MD, MS, Principal Investigator — Yale University
Locations (26):
- United States (26):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California - Davis, Davis, California
  - University of California - Los Angeles, Los Angeles, California
  - University of Colorado - Denver, Denver, Colorado
  - Yale School of Medicine, Department of Neurology, New Haven, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - SUNY Downstate Medical Center, Brooklyn, New York
  - SUNY Buffalo, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Nowak RJ, Coffey CS, Goldstein JM, Dimachkie MM, Benatar M, Kissel JT, Wolfe GI, Burns TM, Freimer ML, Nations S, Granit V, Smith AG, Richman DP, Ciafaloni E, Al-Lozi MT, Sams LA, Quan D, Ubogu E, Pearson B, Sharma A, Yankey JW, Uribe L, Shy M, Amato AA, Conwit R, O'Connor KC, Hafler DA, Cudkowicz ME, Barohn RJ; NeuroNEXT NN103 BeatMG Study Team. Phase 2 Trial of Rituximab in Acetylcholine Receptor Antibody-Positive Generalized Myasthenia Gravis: The BeatMG Study. Neurology. 2022 Jan 25;98(4):e376-e389. doi: 10.1212/WNL.0000000000013121. PMID 34857535
- [Derived] Di Stefano V, Lupica A, Rispoli MG, Di Muzio A, Brighina F, Rodolico C. Rituximab in AChR subtype of myasthenia gravis: systematic review. J Neurol Neurosurg Psychiatry. 2020 Apr;91(4):392-395. doi: 10.1136/jnnp-2019-322606. Epub 2020 Feb 25. PMID 32098874
- [Derived] Hehir MK, Hobson-Webb LD, Benatar M, Barnett C, Silvestri NJ, Howard JF Jr, Howard D, Visser A, Crum BA, Nowak R, Beekman R, Kumar A, Ruzhansky K, Chen IA, Pulley MT, LaBoy SM, Fellman MA, Greene SM, Pasnoor M, Burns TM. Rituximab as treatment for anti-MuSK myasthenia gravis: Multicenter blinded prospective review. Neurology. 2017 Sep 5;89(10):1069-1077. doi: 10.1212/WNL.0000000000004341. Epub 2017 Aug 11. PMID 28801338
- See also: NeuroNEXT Network — http://www.neuronext.org/
- See also: Yale School of Medicine, Department of Neurology — http://medicine.yale.edu/neurology/index.aspx
- See also: National Institutes of Health — http://www.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 68 study participants were consented and assessed for eligibility. 14 participants were ineligible. 2 participants declined. 52 study participants were randomized.
Groups:
- Rituximab: - Treatment group received two cycles of rituximab (375mg/m2 iv), separated by 6 months. Each cycle defined as one infusion per week for four consecutive weeks. For the main study, participants were followed for 52 weeks. Study participants had clinical evaluations performed by a blinded evaluator at baseline and every 4 weeks thereafter.
- Placebo Group: - Placebo group received infusion containing only vehicle components of rituximab solution. Infusion was done in 2 cycles, separated by 6 months. Each cycle defined as one infusion per week for four consecutive weeks. For the main study, participants were followed for 52 weeks. Study participants had clinical evaluations performed by a blinded evaluator at baseline and every 4 weeks thereafter.
Period: Overall Study
Arm/Group | Rituximab | Placebo Group
Started | 25 | 27
No. Completing Study Through Week 52 | 23 | 24
Completed (No. of participants who completed two-cycle rituximab/placebo treatment) | 20 | 23
Not Completed | 5 | 4
Not completed — Adverse Event | 2 | 3
Not completed — Patients who didn't receive 2nd infusion | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: - Placebo group received infusion containing only vehicle components of rituximab solution. Infusion was done in 2 cycles, separated by 6 months. Each cycle defined as one infusion per week for four consecutive weeks. For the main study, participants were followed for 52 weeks. Study participants had clinical evaluations performed by a blinded evaluator at baseline and every 4 weeks thereafter.
- Total: Total of all reporting groups
Arm/Group | Rituximab | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (17.5) | 56.8 (17.0) | 55.1 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 14 | 15 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and ethnicity: Asian | 0 | 1 | 1
  Race and ethnicity: African American | 2 | 9 | 11
  Race and ethnicity: Hispanic | 3 | 2 | 5
  Race and ethnicity: Non-Hispanic white | 20 | 15 | 35
Baseline Prednisone Dose [Mean (Standard Deviation); unit: mg/day] | 23 (11.2) | 21.3 (8.3) | 22.1 (9.7)
Baseline Myasthenia Gravis Composite (MGC) [Mean (Standard Deviation); unit: units on a scale] — The Myasthenia Gravis Composite (MGC) scale consists of test items from the MG-ADL (Myasthenia Gravis Activities of Daily Living) scale and the QMG (Quantitative Myasthenia Gravis Scale) that measure symptoms and signs of MG, with weighted response options. The minimum score is 0, and the maximum score is 50. Higher scores correlate with clinical worsening of the disease.
  units on a scale | 11.1 (6.1) | 8.5 (4.0) | 9.8 (5.2)
Baseline Quantitative Myasthenia Gravis (QMG) [Mean (Standard Deviation); unit: units on a scale] — The Quantitative Myasthenia Gravis Score (QMG) is a commonly used objective outcome measure in myasthenia gravis (MG) comprising 13 items measuring ocular, bulbar, extremity fatigue/strength, and respiratory function (forced vital capacity), each with a possible score from 0 to 3, and a maximum possible of 39 points, where a higher score indicates more severe disease.
  units on a scale | 11.0 (5.1) | 9.2 (3.9) | 10.1 (4.5)
Baseline MG-Activities of Daily Living Score [Mean (Standard Deviation); unit: units on a scale] — This 8 point scale with a maximum score of 24 and a minimum of 0 assesses the subject's ability to perform daily activities and can be performed in approximately 5 minutes. A higher score indicates more severe disease.
  units on a scale | 5.8 (3.6) | 4.0 (3.4) | 4.9 (3.6)
Baseline MG-Quality of Life (MG-QOL) score [Mean (Standard Deviation); unit: units on a scale] — The subject completes the 15-question MG-QOL questionnaire and reports the effect of MG on their quality of life. The MG-QOL should be administered prior to other outcomes evaluations at each visit.The maximum score is 60 and the minimum is 0. A higher score indicates more severe disease.
  units on a scale | 22.7 (14.1) | 17.7 (10.6) | 20.1 (12.5)
Baseline MGFA Clinical Classification Grade [Count of Participants; unit: Participants] — Class I- Any ocular muscle weakness, may have weakness of eye closure, all other muscle strength is normal. Class II - Mild weakness affecting other than ocular muscles, may also have ocular muscle weakness of any severity. Class III - Moderate weakness affecting other than ocular muscles, may also have ocular muscle weakness of any severity. Class IV - Severe weakness affecting other than ocular muscles, may also have ocular muscle weakness of any severity. A higher grade is indicative of a worse outcome.
  Participants
    Class I | 0 | 1 | 1
    Class II | 15 | 16 | 31
    Class III | 9 | 9 | 18
    Class IV | 1 | 1 | 2
Thymectomy [Count of Participants; unit: Participants] | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Steroid Sparing Effect
Description: Percent of subjects that achieve a ≥ 75% reduction in mean daily prednisone dose in the 4 weeks prior to week 52 and have clinical improvement or no significant worsening of symptoms (≤ 2 point increase in MGC score) as compared to 4-week period prior to randomization and initiation of treatment.
Time Frame: 4 weeks prior baseline and 4 weeks prior to week 52
Population: Intention to treat participants
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 25 | 27
Participants | 15 | 15
Statistical Analysis 1: Comparison: Rituximab vs Placebo; This futility design tests the following hypothesis: H0: Rituximab improves outcome by at least 30% compared to placebo (pR - pP ≥ 0.30 - not futile) versus HA: Rituximab does not improve outcome by at least 30% compared to placebo (pR - pP < 0.30 - futile); Test type: Other — A futility (non-superiority) design is a screening tool to identify whether agents should be candidates for phase III trials while minimizing costs/sample size If "futility" is declared, results would imply not cost effective to conduct a future phase III clinical trial If "futility" is not declared, suggests that there could be a clinically meaningful effect - supports exploration in a larger, phase III trial; p = 0.03, Regression, Logistic; Odds Ratio (OR) = 1.14, 90% CI 1-sided [upper limit 2.41]

2. Primary Outcome: Safety:Percentage of Study Participants With Treatment-related Adverse Experiences
Description: Evaluate treatment-Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: 52 weeks
Population: Intention to treat participants
Measure: Count of Participants; unit: Participants
Groups:
- Rituximab: - Treatment group received two cycles of rituximab (375mg/m2 iv), separated by 6 months.Each cycle defined as one infusion per week for four consecutive weeks.For the main study, participants were followed for 52 weeks.Study participants had clinical evaluations performed by a blinded evaluator at baseline and every 4 weeks thereafter.
- Placebo: - Placebo group received infusion containing only vehicle components of rituximab solution. Infusion was done in 2 cycles
  , separated by 6 months. Each cycle defined as one infusion per week for four consecutive weeks. For the main study, participants were followed for 52 weeks. Study participants had clinical evaluations performed by a blinded evaluator at baseline and every 4 weeks thereafter.
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 25 | 27
Participants
  % of participants with treatment related AEs | 19 | 22
  % participants with treatment related SAEs | 6 | 8
Statistical Analysis 1: Comparison: Rituximab vs Placebo; % of study participants with treatment related AEs; Test type: Superiority; p = 0.63, t-test, 2 sided; Odds Ratio (OR) = 0.72, 90% CI 2-sided [0.23 to 2.21]
Statistical Analysis 2: Comparison: Rituximab vs Placebo; % study participants with treatment related SAEs; Test type: Superiority; p = 0.65, t-test, 2 sided; Odds Ratio (OR) = 0.75, 90% CI 2-sided [0.27 to 2.11]

3. Secondary Outcome: Change in Myasthenia Gravis Composite (MGC) Scores From Baseline to Week 52
Description: Evaluate whether there is a trend towards clinical benefit at end of 52 week treatment period, as measured by mean change in the MGC score, an MG-specific clinical outcomes scale used as endpoint in prior MG clinical trials. The Myasthenia Gravis Composite (MGC) scale consists of test items from the MG-ADL (Myasthenia Gravis Activities of Daily Living) scale and the QMG (Quantitative Myasthenia Gravis Scale) that measure symptoms and signs of MG, with weighted response options. The minimum score is 0, and the maximum score is 50. Higher scores correlate with clinical worsening of the disease.
Time Frame: baseline and 52 weeks
Population: Intention to treat participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 25 | 27
score on a scale | -5.7 (7.26) | -4.0 (4.10)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; This objective was assessed longitudinally by comparing the final score at the end of the study to the score obtained at baseline. The outcome was defined as the change from baseline to week 52 in the MGC. This hypothesis was assessed using a linear regression model, adjusted for differences in baseline MGC scores; Test type: Other; p = 0.93, Regression, Linear; Mean Difference (Final Values) = -0.11, 90% CI 1-sided [upper limit 2.02]

4. Secondary Outcome: Change in Quantitative Myasthenia Gravis(QMG) Scores From Baseline to Week 52
Description: Evaluate whether there is a trend towards clinical benefit at end of 52 week treatment period, as measured by the mean change in the QMG score - a specific clinical outcome scale used as endpoint in prior MG clinical trials. The Quantitative Myasthenia Gravis Score (QMG) is a commonly used objective outcome measure in myasthenia gravis (MG) comprising 13 items, each with a possible score from 0 to 3, and a maximum possible of 39 points, where a higher score indicates more severe disease.
Time Frame: baseline and 52 weeks
Population: Intention to treat participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rituximab | Placebo
Number analyzed (Participants) | 25 | 27
score on a scale | -3.95 (5.43) | -1.70 (3.91)
Statistical Analysis 1: Comparison: Rituximab vs Placebo; This objective was assessed longitudinally by comparing the final score at the end of the study to the score obtained at baseline. The outcome was defined as the change from baseline to week 52 in the QMG. This hypothesis was assessed using a linear regression model, adjusted for differences in baseline QMG scores; Test type: Other; p = 0.39, Regression, Linear; Mean Difference (Final Values) = -1.09, 90% CI 1-sided [upper limit 1.03]

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | Rituximab | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/27
Serious Adverse Events (participants affected / at risk) | 9/25 | 14/27
Other Adverse Events (participants affected / at risk) | 25/25 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=25) | Placebo Group (N=27)
Worsening of MG (Nervous system disorders) | 1 (1) | 3 (4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (2)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Micrographic skin surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab (N=25) | Placebo Group (N=27)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 6 (10)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 3 (3) | 8 (9)
Influenza like illness (General disorders) | 3 (4) | 2 (2)
Oedema peripheral (General disorders) | 1 (1) | 2 (3)
Pyrexia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 3 (4)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)
Oral candidiasis (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 2 (3) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 9 (12) | 5 (5)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (5)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Weight increased (Investigations) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 10 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (11)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 4 (5)
Neck pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (9)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 8 (11) | 7 (13)
Paraesthesia (Nervous system disorders) | 0 (0) | 5 (7)
Tremor (Nervous system disorders) | 2 (3) | 3 (4)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Cataract operation (Surgical and medical procedures) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Injection site reaction (General disorders) | 2 (3) | 0 (0)
Fungal skin infection (Infections and infestations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/06/NCT02110706/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT02110706/SAP_001.pdf